CLINICAL TRIAL: NCT00450827
Title: Combination of Targeted I -3F8-Mediated Radioimmunotherapy and Bevacizumab in Patients With Relapsed or Refractory Neuroblastoma: A Phase I Study
Brief Title: Iodine I 131 Monoclonal Antibody 3F8 and Bevacizumab in Treating Patients With Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-072; P30CA008748 (NIH); MSKCC-06072
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Bevacizumab; Filgrastim

ARMS (1):
- Iodine I 131 Monoclonal Antibody 3F8 and Bevacizumab (Experimental): Patients will be administered a therapeutic doses of intravenous (IV) 131I-3F8 given in a single dose per the dose escalation regimen on day 0 of study. This will be followed by blood draws for pharmacokinetic and dosimetry studies and by gamma camera scan, where feasible. Bevacizumab will be administered at a fixed dose of 15mg/kg on days 1 and 15. Thyroid protection is commenced 10 days prior to administration of 131I-3F8 and continued for 28 days after the therapeutic dose of 131I-3F8. ASCR will be carried out if ANC < 500/ul on day 28 (blood radioactivity will be confirmed to be <1 uCi/ml prior to ASCR). ASCR will be carried out sooner in the case of life-threatening infection in the setting of neutropenia (ANC<500). G-CSF can be used to maintain ANC>500/ul but should not be used for 24 hours immediately before and after ASCR. Blood product support will be provided with platelet and red cell transfusions as required.
  Interventions: Biological: bevacizumab; Biological: filgrastim; Procedure: autologous hematopoietic stem cell transplantation; Radiation: iodine I 131 monoclonal antibody 3F8

INTERVENTIONS:
Biological: bevacizumab
Biological: filgrastim
Procedure: autologous hematopoietic stem cell transplantation
Radiation: iodine I 131 monoclonal antibody 3F8

SUMMARY:
RATIONALE: Monoclonal antibodies, such as iodine I 131 monoclonal antibody 3F8 and bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of neuroblastoma by blocking blood flow to the tumor. Giving iodine I 131 monoclonal antibody 3F8 together with bevacizumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of iodine I 131 monoclonal antibody 3F8 when given together with bevacizumab in treating patients with relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of iodine I 131 monoclonal antibody 3F8 (^131I-3F8) and bevacizumab in patients with relapsed or refractory neuroblastoma.
* Determine the hematopoietic recovery after autologous stem cell rescue in patients treated with this regimen.

Secondary

* Determine the clinical response rates in patients treated with this regimen.
* Assess whole body dosimetry for ^131I-3F8.
* Assess tumor targeting of ^131I-3F8 before and after bevacizumab.

OUTLINE: This is a dose-escalation study of iodine I 131 monoclonal antibody 3F8 (^131I-3F8).

Patients receive ^131I-3F8 IV over 20-30 minutes on day 0 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 4 courses. Patients whose blood counts do not recover and whose human antimouse antibody (HAMA) titer < 1,000 U/mL after course 1 receive one dose of ^131I-3F8 alone followed by autologous stem cell rescue (ASCR) and filgrastim (G-CSF). Patients whose blood counts do not recover and whose HAMA titer ≥ 1,000 U/mL after course 1 undergo ASCR followed by G-CSF. Patients whose blood counts recover and whose HAMA titer < 1,000 U/mL after course 1 receive 3 more courses of ^131I-3F8 and bevacizumab in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of ^131I-3F8 and bevacizumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed at 3-4 weeks and then every 3-6 months thereafter.

ELIGIBILITY:
Subject Inclusion Criteria:

* Patients must have the diagnosis of NB in accordance with the International Criteria, i.e., either histopathology (confirmed by the MSKCC Department of Pathology) or BM involvement plus elevated urinary catecholamines.
* Must have a history of tumor progression or recurrence or failure to achieve complete response with standard therapy.
* Patients must have evaluable (microscopic marrow metastasis, MIBG or PET scans) or measurable (CT, MRI) disease.
* Prior Therapy: At least 2 weeks should have elapsed since any biologic therapy. Three weeks should have elapsed since last dose of chemotherapy or radioimmunotherapy.
* Age >1 year and able to cooperate with radiation safety restrictions during therapy period.
* Stem cells: Patients must have an autologous hematopoietic stem cell product cryopreserved and available for re-infusion after MIBG treatment. The minimum dose for hematopoietic stem cells is 2 X106 CD34+ cells/kg.
* Minimum life expectancy of four weeks.
* Signed informed consent indicating awareness of the investigational nature of this program.

Subject Exclusion Criteria:

* Severe major organ toxicity. Renal, cardiac, hepatic, pulmonary, gastrointestinal and neurologic toxicity should all be grade 2 or less (per NCI CTC version 3 criteria). Specifically, serum creatinine should be ≤3 x upper limit of normal (ULN), serum AST and ALT ≤5 x ULN, serum bilirubin ≤ 3 x ULN, LV shortening fraction should be ≥15%.
* Patients with myelosuppression are not excluded if ANC ≥ 500/uL. Platelet count should be > 50,000/ul and hemoglobin should be > 8gm/dl. Patients may receive platelet or red blood cell transfusions to maintain hemoglobin and platelets at clinical appropriate levels.
* Patients with documented chronic non-healing wound, ulcer or bone fracture
* Surgical procedures.
* Patients who have undergone major surgery <28 days prior to beginning therapy with bevacizumab are excluded.
* Patients must be least 24 hours from having after surgical procedures such as placement of central catheter.
* Patients <7days from minor surgeries (e.g. fine needle or core biopsies) and/or the unhealed wounds from these procedures are excluded.
* Patients will be excluded if major surgery (e.g. abdominal or thoracic surgery for resection of tumor) is anticipated during the course of the study.

Known bleeding diathesis or coagulopathy. Patients on anti-coagulants (except for heparin flushes for centra venous catheter maintenance) are excluded.

* Thrombosis: patients must not have had a deep venous or arterial thrombosis (non-central venous catheter related) within the last three months prior to study entry. Patients with cerebrovascular accident or transient ischemic attack within 6 months of therapy are excluded. Patients with history of peripheral vascular disease, myocardial infarction or unstable angina are excluded.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study entry.
* Pulmonary or CNS metastases: pre-therapy CT or MRI of head and chest must be carried out.
* Proteinuria: Urine protein: creatinine ratio ≥ 1.0
* Uncontrolled hypertension.
* HAMA >1000 ELISA units/ml.
* History of allergy to mouse proteins, Chinese hamster ovary cells products or other recombinant human antibodies
* Active serious infections not controlled by antibiotics.
* Pregnant women are excluded for fear of danger to the fetus. Therefore negative pregnancy test is required for all women of child-bearing age, and appropriate contraception is used during the study period.
* Inability or unwillingness to comply with radiation safety procedures or protocol requirements.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shakeel Modak, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Nai-Kong V. Cheung, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States